CLINICAL TRIAL: NCT07327034
Title: A Randomized, Double-blind, Multi-center, Phase 2 Study to Assess the Efficacy and Safety of ABSK-011 Plus Best Supportive Care (BSC) vs. Placebo Plus BSC in Previously Systemically Treated Advanced or Unresectable Hepatocellular Carcinoma Patients With FGF19 Overexpression
Brief Title: ABSK-011+BSC vs. Placebo+BSC in Previously Treated Advanced HCC With FGF19 Overexpression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABSK-011-205
Record Dates: First submitted 2025-11-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; FGF19 overexpression; ABSK-011
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): ABSK-011 plus BSC
  Interventions: Drug: ABSK-011+BSC
- Control arm (Placebo Comparator): Placebo plus BSC
  Interventions: Drug: Placebo+BSC

INTERVENTIONS:
Drug: ABSK-011+BSC — ABSK-011 capsules will be provided and should be taken twice daily, with an interval of approximately 12 hours. The investigational product should be taken with food, with approximately 150 mL of water.
  Arms: Experimental arm
Drug: Placebo+BSC — Placebo capsules will be provided and should be taken twice daily, with an interval of approximately 12 hours. The investigational product should be taken with food, with approximately 150 mL of water.
  Arms: Control arm

SUMMARY:
This is a randomized, double-blind, multicenter, Phase 2 study to evaluate the efficacy and safety of ABSK-011 plus BSC versus placebo plus BSC in advanced or unresectable hepatocellular carcinoma (HCC) patients with FGF19 overexpression who have received prior systemic therapy. Approximately 141 advanced or unresectable HCC patients with FGF19 overexpression who have received prior systemic therapy will be enrolled and randomized to experimental arm or control arm in a 2:1 ratio. Patients will receive assigned study treatment, every 28-day treatment cycle within 1 day of randomization until disease progression, intolerable toxicity, start of new anti-tumor therapy, death, patient refuse to continue treatment, loss to follow-up, or other reasons leading to treatment discontinuation. Immediate BICR review is required for patients with radiographic disease progression as assessed by the investigator. If disease progression is assessed by BICR, the investigator is allowed to unblind after disease progression according to the protocol-specified procedures. After unblinding, patients in the experimental arm, study drug should be discontinued. Patients in the control arm may be transferred to receive ABSK-011 plus BSC after assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patients should be able and willing to comply with study visits and procedures as per protocol.
2. Patients (male or female) ≥ 18 years of age at the time of signing the informed consent form.
3. Patients with advanced or unresectable HCC confirmed histologically/cytologically or clinically according to the American Association for the Study of Liver Diseases (AASLD) criteria (for patients with cirrhosis).
4. Have received at least one prior PD- (L) 1 inhibitor approved as a single agent or in combination for the treatment of HCC and at least one mTKI approved for the treatment of HCC.
5. BCLC stage B(ineligible for local or radical therapy, or relapse or progression of disease after local therapy or radical therapy) or C.
6. Child-Pugh class A.
7. Positive for FGF19 overexpression.
8. At least 1 measurable lesion meeting RECIST v1.1 criteria.
9. ECOG performance status 0 or 1.
10. Life expectancy ≥ 3 months.
11. Adequate control of blood pressure (BP) at screening.
12. Adequate organ function and bone marrow function.
13. Non-surgically sterilized male or female patients of childbearing potential must agree to use reliable contraception for at least 2 weeks prior to randomization until 1 month after the last dose of study treatment.

Exclusion Criteria:

1. Known allergies or hypersensitivity to any component of the investigational product (ABSK-011 or placebo).
2. Previous treatment with selective FGFR4 inhibitors.
3. Known fibrolamellar HCC, sarcomatous HCC, or mixed hepatocellular carcinoma-cholangiocarcinoma.
4. Previous anti-tumor therapy is ≤ 4 weeks from randomization.
5. Major surgery within 4 weeks prior to randomization; or any surgical wound infection, dehiscence, or incomplete healing within 2 weeks prior to randomization; Or major surgery is planned during study treatment.
6. History of second primary malignancies other than HCC within the first 5 years of screening.
7. Liver tumors as a percentage of whole liver ≥ 50% as judged by the investigator.
8. Toxicities caused by prior chemotherapy, radiotherapy, and other anti-tumor therapies (including immunotherapy) did not recover to ≤ Grade 1 CTCAE v5.0.
9. Imaging revealed HCC involving the main portal vein (Vp4), inferior vena cava, superior vena cava, superior mesenteric vein, or heart.
10. Impaired cardiac function or clinically important heart disease.
11. Patients coinfected with HBV and HCV.
12. Known acquired immunodeficiency syndrome (AIDS) -associated disease or tested positive for HIV 1/2 antibodies.
13. Active or documented gastrointestinal bleeding within 6 months prior to screening.
14. Patients with intractable/uncontrolled pleural or pericardial effusion requiring intervention within 2 weeks prior to randomization and clinically significant ascites.
15. Prior or current hepatic encephalopathy (any grade).
16. Presence of meningeal or central nervous system (CNS) metastases.
17. Previous organ transplant and anti-rejection drug therapy indicated.
18. The factors that significantly affect the absorption of oral drugs.
19. Receipt of P-gp transporter inhibitors or moderate, strong inhibitors or inducers of CYP3A4 within 2 weeks prior to randomization.
20. Any serious acute or chronic infection requiring systemic antibacterial, antifungal, or antiviral therapy within 2 weeks prior to randomization.
21. Patient who cannot be assessed by contrast-enhanced CT and/or MRI due to allergy to computed tomography (CT) and/or magnetic resonance imaging (MRI) contrast media or other contraindications.
22. Any other clinically significant comorbidities may affect the patient's health or safety, affect the signing of informed consent, affect protocol compliance, or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR by BICR | through study completion, up to 2 years
  Objective response rate (ORR) assessed by Blinded Independent Central Review (BICR) per RECIST v1.1, defined as the proportion of patients achieving complete response (CR) or partial response (PR). Patients who receive crossover treatment or start a new anti-tumor therapy prior to achieve an objective response (PR or CR) will be considered as non-responders.

SECONDARY OUTCOMES:
PFS | through study completion, , up to 2 years
  Defined as the time (months) from randomization to disease progression or death due to any cause, whichever occurs first.
DOR | through study completion, up to 2 years
  Defined as the time (months) from the first documented objective response to disease progression or death due to any cause, whichever occurs first.
DCR | through study completion, up to 2 years
  Defined as the proportion of patients achieving CR, PR, or SD (meeting the minimum criteria for SD lasting at least 6 weeks).
TTP | through study completion, up to 2 years
  Defined as the time (months) from randomization to disease progression.
TTR | through study completion, up to 2 years
  Defined as time (months) from randomization to first objective response.
OS | through study completion, up to 2 years
  Defined as the time (months) from randomization to death due to any cause.
ORR by investigator | through study completion, up to 2 years
  Objective response rate (ORR) assessed by the investigator per RECIST v1.1, defined as the proportion of patients achieving complete response (CR) or partial response (PR).
Adverse events | through study completion, up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and incidence of adverse events leading to dose interruption, dose reduction, and discontinuation of study treatment.
  Eastern Cooperative Oncology Group (ECOG) performance status (PS), laboratory tests, electrocardiogram (ECG), vital signs, and physical examination and changes from baseline.

OTHER OUTCOMES:
Levels of FGF19 in blood samples | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  Changes in selected PD markers before and after treatment.
Cmax | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  maximum observed concentration
Tmax | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  time to maximum observed concentration
AUC | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  area under the concentration-time curve
t1/2 | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  elimination half-life
Vz/F | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  apparent volume of distribution
CL/F | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  apparent oral clearance
Cmax,ss | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  maximum observed concentration of steady-state
Cmin,ss | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1,Cycle 5 Day 1, End of treatment (each cycle is 28 days)
  minimum observed concentration of steady-state
AUCss | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  area under the concentration-time curve of steady-state
AR | Cycle 1 Day 1, Cycle 1 Day 15 (each cycle is 28 days)
  accumulation rate

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing university cancer hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - General Hospital of Easten Theater Command, Nanjing, Jiangsu
  - Nanjing Tianyinshan Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital with NanJing Medical University, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital ofJining Medical University, Jining, Shandong
  - Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital,Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - TianJin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided